CLINICAL TRIAL: NCT06049303
Title: Effects of Paraffin Wax Bath With Joint Mobilization Technique in Rehabilitation of Post-traumatic Stiff Knee
Brief Title: Paraffin Wax Bath With Joint Mobilization Technique in Post-traumatic Stiff Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0134 Misbah
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Knee Pain Chronic
Keywords: Post-traumatic stiff knee; Range of motion; Pain; Mobilization
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paraffin wax bath therapy and Maitland joint mobilization techniques (Experimental): Paraffin wax bath therapy and Maitland joint mobilization techniques
  Interventions: Other: Paraffin wax bath therapy and Maitland joint mobilization techniques
- Maitland knee joint mobilization (Active Comparator): Maitland knee joint mobilization
  Interventions: Other: Maitland knee joint mobilization

INTERVENTIONS:
Other: Paraffin wax bath therapy and Maitland joint mobilization techniques — In group A Patients will be treated with paraffin wax bath 20 minutes (before any physical therapy treatment)
  * (Apply a few drops of olive oil into the skin of the area. Dip/pour knee joint area into the wax and leave it in for a few seconds until a layer forms over the area. Wait for the wax to dry. Repeat this process until you have at least 10 layers of wax area to be treated.)
  * Joint mobilization technique (8-12 glides at knee joint, mobilization grade-I and grade-II will be used for pain management and relaxation, while grade III for improvement in the PROM at knee joint) will be given 4 times a week for 6 weeks (The patient will be positioned in supine lying with the knee slightly flexed and a prop placed under the distal femur. The stabilizing hand will be used to prop the distal femur and the mobilizing hand is placed over the proximal tibia just below the tibial tuberosity. The mobilization itself will be performed by a force perpendicular to the line of the tibia.)
  Arms: Paraffin wax bath therapy and Maitland joint mobilization techniques
Other: Maitland knee joint mobilization — Group B will have (8-12 glides at knee joint, mobilization grade-I and grade-II will be used for pain management and relaxation, while grade III for improvement in the PROM at knee joint) 4 times a week for 6 weeks.
  Mobilization procedure will be same as above
  Arms: Maitland knee joint mobilization

SUMMARY:
This project will be a Randomized clinical trial conducted to check the effect of paraffin wax bath with joint mobilization technique in rehabilitation of post-traumatic stiff knee joint. Study duration will be of 8 months, convenient sampling was done, subject following eligibility criteria from Jinnah Hospital Lahore, will be randomly allocated in two groups, baseline assessment was done, Group A participants were given baseline treatment along with paraffin wax bath therapy and Maitland knee joint mobilization, Group B participants will be given baseline treatment along with Maitland knee joint mobilization. Assessments will done in 4th week and 8th week via, Numeric pain rating scale, goniometer, western Ontario and McMaster universities osteoarthritis index,4 sessions per week will given, data will analyzed by using SPSS version 25.

DETAILED DESCRIPTION:
Knee stiffness is common problem post traumatically due to process of inhibition often occurs in the early post-injury phase. This leads to the initiation of muscle atrophy within hours of the cessation of normal voluntary muscle activation further; this can result in an increase in the viscosity of synovial fluid within the joint, which provides more resistance to motion. Maitland mobilization aims to reestablish the spinning, gliding and rolling motions of the two joints. Although paraffin bath therapy has various effects such as analgesia, reducing chronic inflammation, and increasing connective tissue elasticity, it is non-invasive and has few side effects. Paraffin wax therapy, combined with exercises and the use of splints, has also been found helpful in restoring the range of movement. The current study is to explore the effect of parrafin wax bath therapy in rehabilitation of posttrumatic stiff knee range of motion, pain and functional status, and emphasize the importance of parrafin wax bath therapy adjunct with mobilization technique in treatment of knee stiffness

ELIGIBILITY:
Inclusion Criteria:

* Age 22-40 yrs.
* Both Male and female
* Fracture of unilateral knee joint.
* Subject with 3-6 month after injury
* Subjects with post traumatic stiffness of knee joint having a minimum of 70º knee flexion

Exclusion Criteria:

* Recent injuries on knee or on adjacent areas.
* Neurological problems
* Subject having polyarthritis, bleeding disorders, tumors, local infection, peripheral vascular disease, leg-length discrepancy of more than one-half inch
* Any non-traumatic cause of fractures
* Non traumatic cause of knee stiffness
* Malignancy

Ages: 22 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
NPRS | 3rd day
  Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain
WOMAC | 3rd day
  Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright, Stiffness (2 items): after first waking and later in the day, Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties.
Goniometer | 3rd day
  A goniometer is an instrument which measures the available range of motion at a joint.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil ur Rehman, Principal Investigator — Riphah International University, Lahore, Pakistan
Locations (1):
- Jinnah Hospital Lahore, Rehab Care, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balasundaram AP, Sreerama Rajan S. Short-term effects of mobilisation with movement in patients with post-traumatic stiffness of the knee joint. J Bodyw Mov Ther. 2018 Apr;22(2):498-501. doi: 10.1016/j.jbmt.2017.06.007. Epub 2017 Jun 15. PMID 29861257
- [Background] Jawade S, Vardharajulu G, Naidu N. Comparison of effectiveness of hold-relax technique and maitlandfs mobilization in improving range of motion in posttraumatic stiffness of knee joint. Journal of Datta Meghe Institute of Medical Sciences University. 2020;15(3):402.
- [Background] Kim SG, Kang JW, Boo JH, Jin DU, Choi SJ, Song GG, Jung JH. Effectiveness of paraffin bath therapy for the symptoms and function of hand diseases: A systematic review and meta-analysis of randomized controlled trials. J Hand Ther. 2023 Jul-Sep;36(3):706-712. doi: 10.1016/j.jht.2022.10.005. Epub 2023 Mar 12. PMID 36914488
- [Background] Riaz HM, Ashraf Cheema S. Paraffin wax bath therapy versus therapeutic ultrasound in management of post burn contractures of small joints of hand. Int J Burns Trauma. 2021 Jun 15;11(3):245-250. eCollection 2021. PMID 34336391
- [Background] Borrell RM, Parker R, Henley EJ, Masley D, Repinecz M. Comparison of in vivo temperatures produced by hydrotherapy, paraffin wax treatment, and Fluidotherapy. Phys Ther. 1980 Oct;60(10):1273-6. doi: 10.1093/ptj/60.10.1273. PMID 7443789
- [Background] Kaneguchi A, Ozawa J, Kawamata S, Yamaoka K. Development of arthrogenic joint contracture as a result of pathological changes in remobilized rat knees. J Orthop Res. 2017 Jul;35(7):1414-1423. doi: 10.1002/jor.23419. Epub 2017 Mar 23. PMID 27601089
- [Background] Simas JM, Kunz RI, Brancalhao RM, Ribeiro Lde F, Bertolini GR. Effects of physical exercise on the cartilage of ovariectomized rats submitted to immobilization. Einstein (Sao Paulo). 2015 Oct-Dec;13(4):574-9. doi: 10.1590/S1679-45082015AO3418. PMID 26761556
- [Background] Rao RV, Balthillaya G, Prabhu A, Kamath A. Immediate effects of Maitland mobilization versus Mulligan Mobilization with Movement in Osteoarthritis knee- A Randomized Crossover trial. J Bodyw Mov Ther. 2018 Jul;22(3):572-579. doi: 10.1016/j.jbmt.2017.09.017. Epub 2017 Sep 28. PMID 30100279
- [Background] Weleslassie GG, Temesgen MH, Alamer A, Tsegay GS, Hailemariam TT, Melese H. Effectiveness of Mobilization with Movement on the Management of Knee Osteoarthritis: A Systematic Review of Randomized Controlled Trials. Pain Res Manag. 2021 May 3;2021:8815682. doi: 10.1155/2021/8815682. eCollection 2021. PMID 34055123
- [Background] Plummer S, Leonard J. Mobilization With Movement as Therapy to Reduce Knee Pain and Increase Knee Range of Motion. J Sport Rehabil. 2022 Jun 20;31(7):950-953. doi: 10.1123/jsr.2021-0294. Print 2022 Sep 1. PMID 35728804